CLINICAL TRIAL: NCT06099353
Title: Effectiveness of Risk Communication Tools and Digital Behaviour Change Platforms to Prevent Cardiovascular Disease in Primary Care: A Cluster Randomised Controlled Trial
Brief Title: Healthy Living With Online suPport & Education for Cardiovascular Disease in the Primary Care Setting
Acronym: HOPE-CVD-GP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Collaborators: National University of Singapore (Other); National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Lee Eng Sing, Assistant Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-2022-928
Record Dates: First submitted 2023-10-18; First posted 2023-10-25 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases (CVD)
Keywords: Primary prevention; Digital health; Genetic risk; Phenotypic risk; Quality of life; Lipids
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Usual Care (No Intervention): * General practitioners' (GPs) usual care for patients.
  * GPs will direct patient participants to a publicly available webpage about managing CVD risk on the Health Promotion Board website.
- Arm 2: Heart Age only (Experimental): * General practitioners' (GPs) usual care for patients.
  * GPs will direct patient participants to a publicly available webpage about managing CVD risk on the Health Promotion Board website.
  * GPs will also show patient participants how to access Heart Age, a risk assessment tool available online and communicate with them their respective Heart Age value.
  Interventions: Behavioral: Heart Age
- Arm 3: Heart Age and Heart Age-HOPE-CVD app (Experimental): * General practitioners' (GPs) usual care for patients.
  * GPs will direct patient participants to a publicly available webpage about managing CVD risk on the Health Promotion Board website.
  * GPs will show patient participants how to access Heart Age, a risk assessment tool available online and communicate with them their respective Heart Age value.
  * GPs will also direct patient participants to download the Heart Age-HOPE- CVD mobile app, an evidence-based behaviour change digital platform.
  Interventions: Behavioral: Heart Age; Behavioral: Heart Age-HOPE-CVD App
- Arm 4: Heart Age, HOPE-CVD app, and genetic risk communication (Experimental): * General practitioners' (GPs) usual care for patients.
  * GPs will direct patient participants to a publicly available webpage about managing CVD risk on the Health Promotion Board website.
  * GPs will show patient participants how to access Heart Age, a risk assessment tool available online and communicate with them their respective Heart Age value.
  * GPs will direct patient participants to download the Heart Age-HOPE- CVD mobile app, an evidence-based behaviour change digital platform.
  * Patient participants will undergo genetic testing from which a genetic risk score for CVD will be estimated. They will be informed which quartile of genetic risk they are at in comparison to the rest of the population. The report also contains information on what this risk means for their chances of developing cardiovascular disease in the future.
  Interventions: Behavioral: Heart Age; Behavioral: Heart Age-HOPE-CVD App; Behavioral: Communication of Genetic Risk Score

INTERVENTIONS:
Behavioral: Heart Age — Heart Age is the phenotypic age based on the risk of the patient participant using a modified tool for CVD risk from the Framingham risk Score. The Heart Age is the age at which an individual would be expected to develop CVD in the next ten years relative to another individual of the same sex and age if all the current CVD risk factors were to be eliminated.
  Arms: Arm 2: Heart Age only; Arm 3: Heart Age and Heart Age-HOPE-CVD app; Arm 4: Heart Age, HOPE-CVD app, and genetic risk communication
Behavioral: Heart Age-HOPE-CVD App — Patient participants will use an online mobile, evidence-based behavioural change psychoeducation application for 24 weeks. New psychoeducational content is released every week. The first seven weeks of the programme seeks to resolve ambivalence about initiating a lifestyle change and increase the readiness and motivation to change. Between Weeks 8 and 15, the platform will support action planning and guide users to execute their preferred self-care behaviour safely and effectively. The remaining nine weeks will provide the user with the skills that will help them with coping and planning to manage relapses and temptations.
  Arms: Arm 3: Heart Age and Heart Age-HOPE-CVD app; Arm 4: Heart Age, HOPE-CVD app, and genetic risk communication
Behavioral: Communication of Genetic Risk Score — General practitioners will draw 3ml of blood from each patient participant for analysis of the patient's genetic risk score of having cardiovascular disease. This genetic risk score will be communicated to the patient, and the communication will include informing patients what cardiovascular disease genetic risk is, what their genetic risk category compared to the population in Singapore is, and what their score means for the future.
  Arms: Arm 4: Heart Age, HOPE-CVD app, and genetic risk communication

SUMMARY:
This pragmatic four-arm (1:1:1:1) parallel cluster randomised controlled trial (cRCT) aims to evaluate the effectiveness of reducing the risk of cardiovascular disease (CVD) through three combinations of interventions for individuals at risk of CVD in the primary care setting in Singapore. These interventions are a) communicating an individual's phenotypic risk of CVD, b) a digital psychoeducation application (Heart Age-HOPE-CVD app) that supports health-promoting behavioural change, and c) communicating an individual's genetic risk of CVD. Our study hypothesis is that the exposure of these three interventions will have additive effects on the primary and secondary objectives.

The primary objective of our study is to evaluate the impact of each intervention arm compared to usual care (Arm 1) on the risk for CVD, using change in low-density lipoprotein cholesterol (LDL) measurements as the outcome measure. The secondary objective is to evaluate the impact of each intervention arm compared to usual care (Arm 1) on the following: (a) individual CVD risk factors (i.e. blood pressure, total cholesterol, high-density lipoprotein, body mass index, smoking status, fasting blood glucose or glycated haemoglobin, diagnosis of diabetes, triglycerides level), (b) risk for CVD (i.e., estimated using the Framingham Risk Score), (c) health-related quality of life and well-being, and (d) practice of health-promoting behaviours.

The Heart Age-HOPE-CVD app is a 6-month interventional programme. Hence, the effects of the interventions will be evaluated after a 6-month period. Patients will be recruited by general practitioners (GPs) at primary care clinics around Singapore. After obtaining informed consent at baseline, patients' data will be collected at four time points: baseline, mid-intervention at week 6, post-intervention health screening at week 24 and post-intervention at week 26. All data collection will be conducted at the primary care clinic, except for mid-intervention data which will be collected via an online form.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-74
* Based in Singapore for the duration of study participation (i.e., 6 months)
* Able to read and understand English
* Have access to and is comfortable using a smartphone
* For patients with diabetes, their LDL has to be at least 2.6 mmol/L
* For patients without diabetes, their LDL has to be at least 3.4 mmol/L

Exclusion Criteria

* Have existing heart disease diagnosis or a prior history of any of the following: Angina, Cardiac arrhythmia, Coronary artery disease, Heart failure, Myocardial infarction, Peripheral vascular disease, Revascularisation, Stroke, Transient ischaemic attack
* Patients diagnosed with chronic kidney disease: i.e., eGFR <60ml/min/1.73㎡ OR uACR ≥ 3mg/mmol (30mg/g) OR uPCR >15mg/mmol (150mg/g)
* Patients with serious mental illness (i.e., require assistance in daily activities due to the mental illness)
* Pregnant or planning to be pregnant in the next six months
* Unable to give informed consent
* Diagnosed with a terminal illness or expected life expectancy of less than 12 months
* Patients with triglyceride levels of ≥ 4.5 mmol/L
* Patients on chemotherapy course during the study or less than one month prior to participating in the study
* Patients on long-term oral steroids
* Patients who are already involved in other HOPE studies (e.g. HOPE-Virtual study)

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in low density lipoprotein | Week 0 and Week 24
  Low-density lipoprotein cholesterol will be measured and compared between the measurements at baseline and post-intervention health screening.

SECONDARY OUTCOMES:
Change in 10-year predicted absolute risk of cardiovascular disease | Week 0 and from Week 24
  Patients' baseline and post-intervention 10-year predicted absolute cardiovascular disease risk will be calculated and compared by a version of the Framingham Risk Score, which is used in the Heart Age algorithm.
  The variables (i.e., age, total cholesterol, high-density lipoprotein cholesterol, diabetes prevalence, smoking status, systolic blood pressure, and prescription of anti-hypertensive medications) needed for this algorithm will be measured or obtained at the baseline and post-intervention health screening visits. These variables will be aggregated into a percentage score ranging from 0-100%, where a higher percentage indicates a higher 10-year predicted absolute risk of CVD. A reduction in the percentage score is a better outcome.
Change in systolic blood pressure | Week 0 and from Week 24
  Systolic blood pressure will be measured and compared between the measurements at baseline and post-intervention health screening visits.
Change in total cholesterol | Week 0 and from Week 24
  Total cholesterol will be measured and compared between the measurements at baseline and post-intervention health screening visits.
Change in high-density lipoprotein cholesterol | Week 0 and from Week 24
  High-density lipoprotein cholesterol will be measured and compared between the measurements at baseline and post-intervention health screening visits.
Change in body mass index | Week 0 and from Week 24
  Body mass index (BMI) will be compared between the measurements at baseline and post-intervention health screening visits. BMI will be calculated by dividing weight in kilograms and the square of height in metres (kg/m2).
Change in smoking habit | Week 0 and from Week 24
  Smoking status will be compared between baseline and post-intervention screening visits. The GP will ask the patient participant if she/he is a smoker at the baseline and post-intervention screening visits, and the GP will collect a "Yes" or "No" response.
Change in fasting blood glucose or glycated haemoglobin measurement | Week 0 and from Week 24
  The fasting blood glucose or glycated haemoglobin will be measured and compared between the measurements at baseline and post-intervention health screening visits.
Change in diagnosis of diabetes | Week 0 and from Week 24
  The diagnosis of diabetes will be compared between baseline and post-intervention screening visits. The GP will ask the patient participant if she/he is a smoker at the baseline and post-intervention screening visits, and the GP will collect a "Yes" or "No" response.
Change in triglycerides | Week 0 and from Week 24
  The triglycerides will be measured and compared between the measurements at baseline and post-intervention health screening visits.
Changes in health-promoting behaviours | Week 0, Week 6, and Week 24
  Health-promoting behaviours will be measured using self-reported questionnaires at baseline, 6 weeks, and 6 months to observe changes over the course of the study. This will be measured using the Readiness for Change questionnaire using a scale of 1 to 40, where a higher score indicates a better outcome.
Change in goal-directed behaviours for living well | Week 0 and from Week 24
  Goal-directed behaviours for living well support a process-based approach to well-being which will be measured and compared between baseline and post-intervention follow-up visits using items in the "EvalUationof goal-diRectedbehaviOurstoPromotewell-beIngandheAlth" scale (Euroia-14). There are 18 items on the Euroia-14 that are separated into four sub-scales (i.e. Self-Affirmation, Social Affiliation, Social Roles and Responsibilities, and Eudemonic). All 18 items are scored between 1 and 4, with a higher score indicating a better outcome.
Change in health-related quality of life | Week 0 and from Week 24
  Health-related quality of life will be assessed and compared between baseline and post-intervention follow-up visits using the items from the validated instrument "Short Form 36 version 2" (SF-36v2).

CONTACTS AND LOCATIONS:
Overall Officials: Eng Sing Lee, Principal Investigator — Nanyang Technological University
Locations (1):
- Lee Kong Chian School of Medicine, NTU, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No